CLINICAL TRIAL: NCT00049075
Title: A Phase II Study of Oral Fludarabine Phosphate in Patients With Previously Untreated B-Cell Chronic Lymphocytic Leukemia
Brief Title: Fludarabine in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL2; CAN-NCIC-CL2 (Other: PDQ); BRLX-304160 (Other: Berlex Study Number); CDR0000257836 (Other: PDQ)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of fludarabine in treating patients who have chronic lymphocytic leukemia that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate (complete and partial) in patients with previously untreated B-cell chronic lymphocytic leukemia treated with oral fludarabine.
* Determine the molecular complete response rate in patients who achieve a clinical or immunophenotypic complete response when treated with this drug.
* Determine the progression-free and treatment-free survival of patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Determine the baseline incidence of defined genetic abnormalities in patients treated with this drug.
* Determine the prognostic and predictive significance of defined genetic abnormalities in patients with respect to response to treatment with this drug.
* Determine the prognostic and predictive significance of immunophenotypic profile of patients with respect to response to treatment with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral fludarabine on days 1-5. Treatment repeats every 28 days for 6-8 courses in the absence of disease progression or unacceptable toxicity. Patients in complete remission after 6 courses do not receive further study therapy.

Patients are followed at 2 months and then every 4 months for 2 years.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of B-cell chronic lymphocytic leukemia (CLL)

  * Previously untreated
  * Rai stage I, II, III, or IV
  * Requiring systemic therapy
* Persistent lymphocytosis of greater than 5,000/mm^3

  * Morphologically mature lymphocytes
* Monoclonal B-cell population

  * CD19/CD5/CD23 positive with kappa or lambda light chain restriction by immunophenotyping
* No other lymphoproliferative disorders including prolymphocytic leukemia, mantle cell lymphoma, progression to aggressive B-cell lymphoma, or Richter's syndrome
* No clinical autoimmune hematologic complication of CLL including Coomb's-positive hemolytic anemia or immune thrombocytopenia

  * Positive Coomb's test allowed if no clinical hemolysis

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST and/or ALT no greater than 2 times ULN

Renal

* Creatinine no greater than 2 times ULN

Other

* Accessible for treatment and follow-up
* No known HIV infection
* No active bacterial, viral, or fungal infection requiring systemic antibiotics
* No conditions requiring corticosteroid therapy
* No history of other malignancies except for the following:

  * Adequately treated nonmelanoma skin cancer
  * Curatively treated carcinoma in situ of the cervix
  * Other solid tumors curatively treated with no evidence of disease within the past 5 years
* No other major medical illness that would preclude study
* No known hypersensitivity to fludarabine or its components
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy including monoclonal antibody therapy
* No concurrent autologous or allogeneic stem cell or bone marrow transplantation

Chemotherapy

* No other concurrent cytotoxic drugs

Endocrine therapy

* No concurrent corticosteroids except inhaled or topical corticosteroids

  * No concurrent corticosteroids for nausea prophylaxis

Radiotherapy

* No prior radiotherapy affecting more than 25% of bone marrow and/or involving the pelvic area
* No concurrent radiotherapy

Surgery

* Not specified

Other

* At least 4 weeks since prior investigational agents
* No other concurrent investigational agents

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2002-08-08 (Actual); Primary Completion 2005-07-22 (Actual); Study Completion 2009-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph M. Meyer, MD, FRCPC, Study Chair — Margaret and Charles Juravinski Cancer Centre
Locations (34):
- Canada (32):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Providence Health Care - Vancouver, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Durham Regional Cancer Centre at Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Algoma Reginal Cancer Program at Sault Area Hospital, Sault Ste. Marie, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - St. Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital - Weston, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Hopital de L'Enfant Jesus, Québec, Quebec
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- France (2):
  - Centre Jean Bernard, Le Mans
  - Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shustik C, Turner AR, Desjardins P, Fernandez L, Rubin S, Larratt L, Duncan AM, Rizi D, Sadura A, Shepherd L, Li D, Rassenti L, Kipps T. Oral fludarabine in untreated patients with B-cell chronic lymphocytic leukemia. Leukemia. 2010 Jan;24(1):237-9. doi: 10.1038/leu.2009.205. Epub 2009 Oct 8. No abstract available. PMID 19812607